CLINICAL TRIAL: NCT02573883
Title: A Randomized Trial of Clobetasol Propionate Versus Fractionated CO2 Laser for the Treatment of Lichen Sclerosus (CuRLS)
Brief Title: Clobetasol Propionate Versus Fractionated Carbon Dioxide Laser for the Treatment of Lichen Sclerosus
Acronym: CuRLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-154
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Vulva; Lichen Sclerosus; Fractionated Carbon Dioxide Laser; Mona Lisa Laser; Clobetasol Propionate; Vulvodynia
MeSH Terms: conditions — Vulvar Lichen Sclerosus; Lichen Sclerosus et Atrophicus; Vulvodynia | interventions — Clobetasol; Ointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prior Clobetasol Exposure (Experimental): Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Interventions: Device: Fractionated Carbon Dioxide Laser; Drug: Clobetasol Propionate 0.05% ointment
- No Prior Clobetasol Exposure (Active Comparator): Patients with biopsy proven lichen sclerosus never previously treated with clobetasol propionate.
  Interventions: Device: Fractionated Carbon Dioxide Laser; Drug: Clobetasol Propionate 0.05% ointment

INTERVENTIONS:
Device: Fractionated Carbon Dioxide Laser — Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart.
  Other Names: SmartXide -V2-LR system; Mona Lisa Laser
Drug: Clobetasol Propionate 0.05% ointment — Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment.
  Other Names: Temovate Propionate 0.05% ointment

SUMMARY:
This study is being done to compare the effects, good and bad, of fractionated CO2 laser treatment and clobetasol propionate .05% ointment on vulvar lichen sclerosus.

DETAILED DESCRIPTION:
Vulvar lichen sclerosus (LS) is a well-characterized dermatosis resulting in labial atrophy, synechiae and introital narrowing and can often cause dyspareunia, itching and co-existent vulvar pain. Biopsy is necessary to confirm the clinical diagnosis and the mainstay of treatment usually consists of topical steroid therapy (Chi). Clobetasol propionate and mometasone furoate are potent topical steroids that have long been considered gold-standard treatment for vulvar lichen sclerosus and work through anti-inflammatory, anti-mitotic, and immunosuppressive effects. One of the complications of long-term steroid use, however, is potential thinning of the vulvar skin, therefore limiting long-term use. Clobetasol propionate has a range of efficacy from 61-91% depending on the selected outcome criteria.

The vulvovaginal SmartXide -V2-LR laser system by DEKA (Calezano, Italy) is a fractionated C02 laser with maximum 40 Watt power and laser energy emission at 10,600 nanometer wavelength which is mainly absorbed by water in the underlying tissue (Salvatore). The SmartXide-V2-LR system was first introduced in 2009 with DOT therapy distributing fractioned CO2 laser in small spots of 200 microns to the vulvar skin or vaginal epithelium, resulting in a portion of the skin remaining intact with less tissue destruction and faster healing (Salvatore). The device is cleared by the US Food and Drug Administration (FDA) for incision, excision, ablation, and coagulation of gynecologic soft tissues. The fractioned therapy has been shown to stimulate fibroblastic growth through activation and biosynthesis of collagen and restoration of the extracellular matrix with collagen fibers.

Very little is known about long-term effects of fractionated C02 laser therapy use in the vulva or vagina, although the treatment is widely accepted in plastic and cosmetic surgery and dermatology. Increased marketing for laser vaginal rejuvenation has spawned a proprietary female genital cosmetic surgery industry in the US with very limited published outcome data. SmartXide -V2-LR has some established outcome data for treatment of genitourinary syndrome of menopause (GSM), also known as vulvovaginal atrophy (Salvatore).

The purpose of this study is to compare the safety and efficacy of clobetasol propionate .05% ointment to fractionated CO2 laser procedure for the treatment of vulvar lichen sclerosus. Women presenting to the urogynecology clinic will be screened for lichen sclerosus. Vulvar biopsy will be performed for confirmation, and, if eligible, the patient will be consented to undergo baseline questionnaires, photodocumentation of vulvar lesions and randomization. A minimum of 2 weeks are required from the time of biopsy to treatment. Patient will be randomized to monthly LASER treatment for 3 months or topical STEROID therapy (clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) in a 1:1 ratio using a computer generated randomization schedule. Because of the nature of the treatment, it will not be possible to blind patients but the assessor will be blinded to the intervention. Patients may have used clobetasol propionate in past, but must complete 8 week wash out period.

Patient questionnaires include multiple validated scales and surveys to provided reproducible measures of vulvar symptoms as primary and secondary outcomes. Questionnaires will be completed at the intake visit, repeated at 6 month and one year follow up. The investigators expect improved subjective and objective results in the LASER group at 6 months compared with the STEROID group. At 6 months, participants are giving the option to crossover to receive the other treatment arm if desired due to continued symptoms. All groups are followed to 12 months for comparison.

Sample size calculations were conducted using the absolute change in the Skindex 29 as the primary end point. Out study will reach 80% power to detect a mean difference of 16 points on the Skindex 29 (sd=22 for both groups) between the study groups with 25 patients in each group, or 50 in total based on a one-sided two-sample t-test with alpha=0.05 (He). By accounting for 10% attrition, the investigators propose to recruit 56 patients to the study to be randomized with a 1:1 ratio to each group, with a blocked component for those who used tropical clobetasol in the past.

Data will be entered into a secure RedCAPS Database which provides complete auditing for data management processes. De-identified backup data will be kept in locked files at the participating site. Plans for publication will be handled by the investigators at MedStar Washington Hospital Center and will adhere to publication policies. All personnel with access to data collected have completed the Program for Ethics Education in Research training with the appropriate HIPAA certification.

Patients will not be compensated for travel and may be accountable for some medical bills for office visits. Study location is Medstar Lafayette Office 1133 21st St NW, Washington, DC 20036.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven symptomatic vulvar lichen sclerosus
* Ability to understand the study, accept randomization and logistically follow-up with scheduled visits
* English Speaking

Exclusion Criteria:

* Known vulvar malignancy
* Pregnancy or planning pregnancy or less than 3 months postpartum
* Premenopausal
* Current or prior diagnosis of any gynecologic malignancy
* Previous pelvic radiation therapy
* Allergy to topical steroid
* Active Urinary Tract Infection (UTI), vulvar infection (candida, herpes, bacterial vaginosis, trichomoniasis or other infection)
* Pelvic organ prolapse > than Stage 2
* Treatment with systemic immunomodulators, topical calcineurin inhibitors (tacrolimus, pimecrolimus), or vaginal hormonal or vulvar topical steroid use within 2 months of enrollment
* History of transvaginal mesh implant (excluding sling or sacrocolpopexy mesh)
* IUD (Intrauterine Device)
* Skindex-29 overall score <21, below mildly impaired health related quality of life threshold

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Iglesia, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center Lafayette Office, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Chi CC, Kirtschig G, Baldo M, Brackenbury F, Lewis F, Wojnarowska F. Topical interventions for genital lichen sclerosus. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD008240. doi: 10.1002/14651858.CD008240.pub2. PMID 22161424
- [Background] Salvatore S, Nappi RE, Zerbinati N, Calligaro A, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. A 12-week treatment with fractional CO2 laser for vulvovaginal atrophy: a pilot study. Climacteric. 2014 Aug;17(4):363-9. doi: 10.3109/13697137.2014.899347. Epub 2014 Jun 5. PMID 24605832
- [Background] He Z, Lu C, Chren MM, Zhang Z, Li Y, Ni X, Buchtel V HA, Ryan PF, Li GZ. Development and psychometric validation of the Chinese version of Skindex-29 and Skindex-16. Health Qual Life Outcomes. 2014 Dec 24;12:190. doi: 10.1186/s12955-014-0190-4. PMID 25539748
- [Derived] Burkett LS, Siddique M, Zeymo A, Brunn EA, Gutman RE, Park AJ, Iglesia CB. Clobetasol Compared With Fractionated Carbon Dioxide Laser for Lichen Sclerosus: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):968-978. doi: 10.1097/AOG.0000000000004332. PMID 33957642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from urogynecologic and gynecology academic center office visits with vulvar biopsy-proven lichen sclerosus. Patients underwent block randomization with a 1:1 ratios, with stratification for participants based on prior clobetasol use. Participates stayed in randomized group until six months when they had the option to crossover into other treatment group and receive that treatment or continue to 12 months with current treatment.
Groups:
- Clobetasol Propionate- No Crossover: Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment then as need. Participants did not cross over.
- Fractionated Carbon Dioxide Laser- No Crossover: Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart. Then no further treatment.
- Clobetasol Propionate to Laser Crossover: Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment then as need. Participants choose to crossover to Fractionated Carbon Dioxide Laser at six months because symptoms had not resolved.
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart.
- Fractionated Carbon Dioxide Laser to Clobetasol Crossover: Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart. Then patients choose to crossover to the Clobetasol Propionate Treatment at six months due to continued symptoms.
  Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment then as need.
Period: Six Month Follow Up
Arm/Group | Clobetasol Propionate- No Crossover | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Started | 25 | 27 | 0 | 0
Completed | 24 | 27 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: One Year Follow Up
Arm/Group | Clobetasol Propionate- No Crossover | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Started | 13 | 17 | 11 | 10
Completed | 11 | 16 | 11 | 10
Not Completed | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fractionated Carbon Dioxide Laser: Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart.
- Clobetasol Propionate: Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment
- Total: Total of all reporting groups
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (11) | 61.5 (8.9) | 64.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 23 | 17 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52
Prior Clobetasol Exposure [Count of Participants; unit: Participants] | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in SkinDEX-29 Score
Description: The Skindex-29 is a validated questionnaire for assessing acute dermatologic symptoms over a 4-week period. The Skindex-29 is a 29 question version of the original SkinDEX questionnaire. Total numeric score is reported ranging from 0-100. Scores reported as a change between six months and baseline with more negative scores indicating greater improvement in symptoms (better outcome).
Time Frame: Change from baseline score to score at six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
score on a scale | -16.83 (18.09) | -5.92 (5.81)
Statistical Analysis 1: Comparison: Fractionated Carbon Dioxide Laser vs Clobetasol Propionate; Test type: Superiority; p = 0.007, t-test, 2 sided

2. Secondary Outcome: Change in Subjective Vulvovaginal Symptoms Questionnaire (VSQ)
Description: Subjective measure of vulvar symptoms of itching, burning, dyspareunia of Lichen Sclerosus. VSQ is a 21-item instrument and scores range from 0 to 20 with increased scores indicating increased vulvovaginal symptom bother. The change in VSQ is reported with more negative scores indicating greater improvement.
Time Frame: Baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
score on a scale | -3.92 (4.12) | -0.58 (5.11)
Statistical Analysis 1: Comparison: Fractionated Carbon Dioxide Laser vs Clobetasol Propionate; Test type: Superiority; p = 0.014, t-test, 2 sided

3. Secondary Outcome: Change in Subjective Vulvovaginal Symptoms Questionnaire (VSQ)
Description: as for outcome 2
Time Frame: Six month to one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
score on a scale | 0.44 (4.43) | 0.3 (2.41) | -1.82 (3.66) | -2.9 (3.98)

4. Secondary Outcome: Number of Participants Considered Satisfied as Assessed by Health Related Quality of Life (HRQOL) Score
Description: Patient global impression of satisfaction total score on visual analog scale (very satisfied or satisfied) ranging from 1-5 with higher scores indicating greater satisfaction.
Time Frame: Six months from treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
Participants | 21 | 9
Statistical Analysis 1: Comparison: Fractionated Carbon Dioxide Laser vs Clobetasol Propionate; Test type: Superiority; p = 0.011, Chi-squared

5. Secondary Outcome: Number of Participants Considered Satisfied as Assessed by Health Related Quality of Life (HRQOL) Score
Description: as for outcome 4
Time Frame: 1 year from treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
Participants | 14 | 4 | 9 | 10

6. Secondary Outcome: Change Vaginal Health Index (VHI) Score
Description: The Vaginal Health Index is a five item scale with scores ranging from 5-25 with lower scores indicating greater urogenital atrophy. The change in VHI is express with more negative scores indicating greater improvement between study time points.
Time Frame: Baseline to 6 months after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
score on a scale | 1.92 (4.34) | -0.43 (3.62)
Statistical Analysis 1: Comparison: Fractionated Carbon Dioxide Laser vs Clobetasol Propionate; Test type: Superiority; p = 0.46, t-test, 2 sided

7. Secondary Outcome: Change Vaginal Health Index (VHI) Score
Description: as for outcome 6
Time Frame: Six month to one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
score on a scale | -2.86 (4.37) | 1.44 (4.45) | 1.73 (2.83) | 1.3 (4.3)

8. Secondary Outcome: Change Vulvar Symptom Visual Analog Scale (VAS) Score
Description: Patient subjective scale of symptoms of Lichen Sclerosus. Each item scaled 0-10 with greater severity of symptoms indicated by higher score. Results expressed as change with more negative values indicating greater improvement.
Time Frame: Baseline to 6 months after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
score on a scale
  Itching | -3.26 (3.75) | -1.83 (2.75)
  Burning | -2.78 (3.76) | -1.00 (3.21)
  Irritation | -4.15 (4.04) | -1.32 (2.84)
  Pain with sex | -0.69 (2.95) | -0.14 (1.35)
  Tearing of vulvar skin | -1.77 (3.55) | -1.32 (4.07)
  Dysuria | -2.11 (3.47) | -0.78 (2.37)
  Pain defecation | -1.11 (2.83) | -0.78 (2.67)

9. Secondary Outcome: Change Vulvar Symptom Visual Analog Scale (VAS) Score
Description: Patient subjective scale of symptoms of Lichen Sclerosus. Each item scaled 0-10 with greater severity of symptoms indicated by higher score. Results expressed as change with more negative values indicating greater improvement in symptoms (better outcome).
Time Frame: Six months to one year after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
score on a scale
  Itching | -0.8 (3.76) | -0.1 (3.03) | -1.82 (3.06) | 0.89 (4.76)
  Burning | -0.73 (3.43) | -1.5 (3.87) | -0.73 (4.45) | -0.9 (2.6)
  Irritation or tearing | -0.38 (4.03) | -1 (3.54) | -1.64 (2.69) | 0.67 (3.71)
  Pain with sex | -1.12 (4.26) | 0 (0) | -1.62 (3.25) | -2 (4)
  Tearing of vulvar skin | -0.14 (3.8) | -0.8 (2.66) | -2.12 (3.14) | -0.22 (1.99)
  Dysuria | -0.5 (4.77) | -0.2 (3.97) | -1.27 (2.94) | -0.4 (0.84)
  Painful defecation | 0 (3.21) | -0.57 (3.98) | -0.09 (1.38) | -0.89 (1.36)

10. Secondary Outcome: Change SkinDEX-29 Score
Description: The Skindex-29 is a validated questionnaire for assessing acute dermatologic symptoms over a 4-week period. The Skindex-29 is a 29 question version of the original SkinDEX questionnaire. Total numeric score is reported ranging from 0-100. Scores reported as a change between six months and baseline with more negative scores indicating greater improvement.
Time Frame: Six months to one year from treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
score on a scale | -0.78 (25.94) | -7.05 (22.13) | -10.23 (17.53) | -1.52 (11)

11. Secondary Outcome: Change Objective Provider VAS Visual Analog Scale
Description: Provider scored objective appearance of vulvar Lichen Sclerosus. Each item scaled 0-10 with greater severity of appearance indicated by higher score. Results expressed as change with more negative values indicating greater improvement.
Time Frame: Baseline to Six months from treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
score on a scale
  White Plaque | -1.81 (1.70) | -1.3 (1.96)
  Cigarette Paper | -2.58 (1.92) | -1.5 (1.9)
  Introital Narrowing | -1.73 (2.82) | -0.70 (2.16)
  Perianal Involvement | -0.73 (3.49) | -1.77 (3.35)
  Loss of Labial Minora | -0.96 (2.44) | -0.78 (2.26)
  Fusion of Labia Minora | -0.5 (2.5) | 0.35 (2.92)
  Phimosis | -1.28 (2.3) | 0.22 (2.04)
  Fissure | -2.12 (2.4) | -1.78 (2.41)
  Erosion | -2.08 (2.86) | -0.57 (1.88)

12. Secondary Outcome: Change Objective Provider VAS Visual Analog Scale
Description: as for outcome 11
Time Frame: Six months to One Year from treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
score on a scale
  White Plaque | -0.71 (3.29) | -1.25 (1.49) | -0.27 (2.24) | -0.22 (1.45)
  Cigarette Paper | 0.07 (3.1) | 0.38 (1.6) | -0.45 (1.81) | -0.2 (1.48)
  Introital Narrowing | 0 (2.6) | 0.88 (2.53) | -0.18 (0.52) | -0.1 (2.42)
  Perianal Involvement | -0.77 (4.07) | 0.29 (1.7) | 0.64 (4.7) | -1.4 (1.9)
  Loss of Labial Minora | 0.5 (2.9) | -0.5 (1.69) | 0.73 (2.8) | 1.2 (2.9)
  Fusion of Labia Minora | 0.14 (2.54) | -0.25 (1.91) | -1.09 (2.59) | -1 (2.83)
  Phimosis | 1.43 (2.21) | -0.5 (1.69) | -0.18 (1.66) | 0.2 (2.53)
  Fissure | 0.07 (2.53) | 0.62 (1.06) | -0.45 (2.62) | -1.4 (2.32)
  Erosion | 1 (2.8) | 0.12 (0.35) | -0.36 (1.03) | -0.6 (1.9)

13. Secondary Outcome: Number of Patients With Adverse Outcomes
Description: Total number for adverse outcomes (of any severity) to include description of pain, infection, de novo or worsening dyspareunia, contact dermatitis and burns from treatment
Time Frame: Six Month to One Year from treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Carbon Dioxide Laser- No Crossover | Clobetasol Propionate- No Crossover | Clobetasol Propionate to Laser Crossover | Fractionated Carbon Dioxide Laser to Clobetasol Crossover
Number analyzed (Participants) | 16 | 11 | 11 | 10
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Patients With Adverse Outcomes
Description: as for outcome 13
Time Frame: 12 Weeks to Six months from treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
Participants | 0 | 0

15. Secondary Outcome: Number of Patients With Adverse Outcomes
Description: as for outcome 13
Time Frame: 12 Weeks from treatment
Population: Please see adverse events section for description of adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Carbon Dioxide Laser | Clobetasol Propionate
Number analyzed (Participants) | 27 | 24
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 12 weeks, six months, and one year post treatment
Groups:
- Clobetasol Propionate- 0-6 Months: Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment then as need.
- Fractionated Carbon Dioxide Laser- 0-6 Months: Patients with biopsy proven lichen sclerosus previously treated with clobetasol propionate
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart.
- Clobetasol Propionate to Laser Crossover 6-12 Months: Participants previously in the Clobetasol Propionate 0.05% ointment group. Participants choose to crossover to Fractionated Carbon Dioxide Laser at six months because symptoms had not resolved.
  Fractionated Carbon Dioxide Laser: Vulvar lichen sclerosis will be treated except for the clitoris glans and clitoral hood which will be spared with at least 5mm margin. The procedure will be performed in the outpatient clinic at the National Center for Advanced Pelvic Surgery at MedStar Washington Hospital Center Lafayette Office, 1133 21st St NW, Washington, DC 20036, and include 3 sessions, 4 weeks apart.
- Fractionated Carbon Dioxide Laser to Clobetasol Crossover 6-12 Months: Participants previously in the Fractionated Carbon Dioxide Laser group choose to crossover to the Clobetasol Propionate Treatment at six months due to continued symptoms.
  Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment nightly for one month then three times weekly for 2 additional months) for a total of three months of treatment then as need.
- Clobetasol Propionate - No Crossover 6-12 Months: Clobetasol Propionate 0.05% ointment Topical Steroid therapy (Clobetasol propionate .05% ointment continued as need. No Crossover.
- Fractionated Carbon Dioxide Laser- No Crossover 6-12 Months: Participants previoulsly treated with Fractionated Carbon Dioxide Laser choose to not undergo any further treatment.
Arm/Group | Clobetasol Propionate- 0-6 Months | Fractionated Carbon Dioxide Laser- 0-6 Months | Clobetasol Propionate to Laser Crossover 6-12 Months | Fractionated Carbon Dioxide Laser to Clobetasol Crossover 6-12 Months | Clobetasol Propionate - No Crossover 6-12 Months | Fractionated Carbon Dioxide Laser- No Crossover 6-12 Months
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/11 | 0/10 | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/11 | 0/10 | 0/11 | 0/16
Other Adverse Events (participants affected / at risk) | 1/27 | 1/24 | 0/11 | 0/10 | 0/11 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate- 0-6 Months (N=27) | Fractionated Carbon Dioxide Laser- 0-6 Months (N=24) | Clobetasol Propionate to Laser Crossover 6-12 Months (N=11) | Fractionated Carbon Dioxide Laser to Clobetasol Crossover 6-12 Months (N=10) | Clobetasol Propionate - No Crossover 6-12 Months (N=11) | Fractionated Carbon Dioxide Laser- No Crossover 6-12 Months (N=16)
minor burning and blistering at treatment site (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — adverse event was minor burning and blistering at laser site
Activation Genital Herpes (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — adverse event was activation of genital herpes one week after starting steroid

LIMITATIONS AND CAVEATS:
The study was unblinded for patients and evaluators and only performed at a single center. The steroid group had more non-compliant patients (25% vs 4%). We limited our investigation to only postmenopausal women Further research using placebo and sham lasers for treatment blinding is needed. Patients previously using topical vaginal estrogen were continued on prior treatment, groups were not stratified based on estrogen exposure, however there where equal numbers between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02573883/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02573883/ICF_001.pdf